CLINICAL TRIAL: NCT00894868
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effect of 52 Weeks Treatment With Vildagliptin on Left Ventricular Function in Patients With Type 2 Diabetes and Congestive Heart Failure
Brief Title: Effect of Vildagliptin on Left Ventricular Function in Patients With Type 2 Diabetes and Congestive Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A23118; 2008-005012-41 (EudraCT Number)
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2014-04

CONDITIONS: Congestive Heart Failure; Type II Diabetes Mellitus
Keywords: Congestive Heart Failure; CHF, vildagliptin; metabolic disease; cardiovascular disease; T2DM
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Metabolic Diseases; Cardiovascular Diseases | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: vildagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo of vildagliptin

INTERVENTIONS:
Drug: vildagliptin
  Arms: Vildagliptin
Drug: placebo of vildagliptin
  Arms: Placebo

SUMMARY:
This study will assess the effect of vildagliptin on left ventricular function in patients with type 2 diabetes and congestive heart failure (NYHA Class I-III). Effect on HbA1c and overall safety and tolerability will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM, diagnosed at least 3 months prior to Visit 1
* CHF (NYHA Class I, Class II, or Class III) at Visit 1
* LVEF < 40%

Exclusion Criteria:

* Pregnant or lactating female
* FPG ≥ 270 mg/dL (≥15 mmol/L)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of vildagliptin on left ventricular function in patients with T2DM and CHF (NYHA class I-III) by showing that vildagliptin is at least not inferior to placebo with respect to change in left ventricular ejection fraction (LVEF). | 52 weeks

SECONDARY OUTCOMES:
To evaluate the overall safety of vildagliptin versus placebo in patients with T2DM and CHF (NYHA class I - III) over 52 weeks of treatment with special regard to signs and symptoms of heart failure. | 52 weeks
To evaluate the efficacy of vildagliptin in patients with T2DM and CHF (NYHA class I-III) by assessing the HbA1c reduction with vildagliptin compared to placebo after 16 weeks of treatment. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (80):
- Czechia (7):
  - Novartis Investigative Site, Benešov, Czech Republic
  - Novartis Investigative Site, Havířov, Czech Republic
  - Novartis Investigative Site, Litomyšl, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Prague, CZE
  - Novartis Investigative Site, Broumov
  - Novartis Investigative Site, Pardubice
- Denmark (6):
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Copenhagen S
  - Novartis Investigative Site, Frederiksberg
  - Novartis Investigative Site, Hellerup
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Slagelse
- Estonia (3):
  - Novartis Investigative Site, Pärnu
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Germany (7):
  - Novartis Investigative Site, Alsdorf
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Kamp-Lintfort
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Senden
- Greece (3):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Chios
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Guatemala City, Guatemala
- India (13):
  - Novartis Investigative Site, Secunderabad, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Indore, Madhya Pradesh
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
- Italy (8):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Passirana Di Rho, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Mercato San Severino, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Novara
- Latvia (2):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Preiļi
- Lithuania (3):
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Kłodzko
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Romania (4):
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Baia Mare, Maramureş
  - Novartis Investigative Site, Brasov
- Russia (11):
  - Novartis Investigative Site, Kaliningrad
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (7):
  - Novartis Investigative Site, Dunajská Streda, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Modava Nad Bodvou

REFERENCES:
- [Derived] McMurray JJV, Ponikowski P, Bolli GB, Lukashevich V, Kozlovski P, Kothny W, Lewsey JD, Krum H; VIVIDD Trial Committees and Investigators. Effects of Vildagliptin on Ventricular Function in Patients With Type 2 Diabetes Mellitus and Heart Failure: A Randomized Placebo-Controlled Trial. JACC Heart Fail. 2018 Jan;6(1):8-17. doi: 10.1016/j.jchf.2017.08.004. Epub 2017 Oct 11. PMID 29032139
- See also: Results for CLAF237A23118 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9563